CLINICAL TRIAL: NCT02234856
Title: Evaluation of Laparoscopic Hysterectomy Simulator to Improve Cognitive Surgical Knowledge of Obstetrics and Gynecology Trainees
Brief Title: Evaluation of Laparoscopic Hysterectomy Simulator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 30509
Record Dates: First submitted 2014-08-06; First posted 2014-09-09 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Evaluation of Laparoscopic Hysterectomy Simulator
Keywords: Hysterectomy; Laparoscopy; Surgical assessment; Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional residency training (No Intervention): no intervention
- Laparoscopic Hysterectomy trainer (Experimental): Intervention: An educational video and web-based e-module will be created. The final product will be reviewed by the expert contributors. Once approved, these tools will be showcased to a voluntary focus group of Obstetrics and Gynecology residents at the University of Toronto. A quantitative assessment of effectiveness of this tool will be performed through the use of pre- and post-tests of knowledge. A qualitative needs assessment will also be performed using post-viewing surveys. If found to be effective, this educational tool will be incorporated in the University of Toronto Obstetrics and Gynecology residency curriculum.
  Interventions: Procedure: Laparoscopic Hysterectomy trainer

INTERVENTIONS:
Procedure: Laparoscopic Hysterectomy trainer — In order to increase comfort level amongst Gynecologists, we aim to identify verbal and non-verbal components of teaching TLH through interview and video recordings. Utilizing qualitative analysis of common themes, we will develop an educational video and web-based e-module to be used by Gynecology residents and surgeons. We will also use a combination of quantitative pre- and post-tests and qualitative surveys to assess the effectiveness of such a training tool. Ultimately, the project aims to create a robust tool that can be implemented in Gynecology residencies.
  Arms: Laparoscopic Hysterectomy trainer

SUMMARY:
This study aims to test the validity of a new educational tool in the form of a computer based video surgical simulator, that may be used to enhance the current teaching method of how to perform a hysterectomy.

DETAILED DESCRIPTION:
Ensuring the surgical competence of trainees is mandatory for all surgical residency programs, yet most evaluations of graduating residents are based on observation and subjective feedback. We have developed a computer based video surgical simulator to facilitate cognitive knowledge of the step-by-step process needed to perform a laparoscopic hysterectomy, learn essential pelvic anatomy and avoid surgical complications. Studies have shown that when trainees already have the cognitive knowledge of how to perform a procedure, they can focus more on learning surgical technique and how to minimize surgical complications. Laparoscopy is becoming the standard of surgical care for gynecologic patients. The benefits of minimally invasive surgery include reduced postoperative pain, shorter hospitalization, less scarring, quicker return to normal activities, preservation of immune response, and fewer long-term problems such as adhesions or incisional hernia. The current challenge in surgical education is how to produce competent surgeons who are skilled to perform and integrate the multiple advances in surgical technology. Surgical competency involves proficiency in technical skills, decision-making (preoperative, operative, and postoperative), and team performance all of which require knowledge and communication skills. The increasing complexity of surgery and the requirements for mastery at laparotomy, laparoscopy, and endoscopy reduces the feasibility of the traditional "see one, do one, teach one" model of surgical education. Lack of training is considered a major barrier to performing laparoscopic surgery. Alternative training modalities are required to acquire the necessary surgical skills for laparoscopy. Although there is a transfer of skills and knowledge to the trainee by the time of graduation, current training programs have not been designed in a validated, effective, and competency-based manner. A successful laparoscopic curriculum should incorporate a cognitive component in addition to the manual skills component. Although the benefit of simulators as a method of surgical education has been validated, comprehensive curriculum development is lacking. Most recently, Zevin et al. (2012) conducted a Delphi consensus involving international experts in surgical education on the principles for design, validation and implementation of a simulation-based surgical training curriculum. The main components of the final framework included predevelopment analysis; cognitive, psychomotor, and team-based training; curriculum validation, evaluation, and improvement; and maintenance of training. They have produced a framework that is based on the broad principles of educational theory that can be applied to any surgical specialty. Several authors have emphasized the importance of cognitive teaching in a comprehensive surgical skills training curriculum. Learning begins with the acquisition of procedure-specific knowledge. Categories include pre-procedure assessment and preparation; anatomic knowledge; safety and limitations of specific instruments; ergonomics; and post-procedure management. A cognitive curriculum can include reading materials in the form of text books or journal articles as well as procedural video tutorials. The cognitive component should be studied by the trainee before technical skills training and should be followed by satisfactory performance on a paper-based test of knowledge or a mock operative note dictation. Teaching about errors commonly associated with the procedure should be included so that trainees can anticipate or avoid them in the future, and recognize and manage them if they occur. The purpose of this research study is to test the validity of a new educational tool as an enhancement to the current teaching method of how to perform a hysterectomy. Should our data substantiate our hypothesis, that cognitive function of surgical trainees will be enhanced by use of the trainer, then the tool will be able to be utilized as a new, advanced, creative tool for teaching how to perform a hysterectomy. This tool might then be able to be utilized to advance the teaching of many other surgical procedures to residents in many different surgical programs.

ELIGIBILITY:
Inclusion Criteria:

* Faculty in the Department of Ob-Gyn
* Experienced OBGYN surgeons
* Residents in the Department of Ob-Gyn

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Number of residents using validation tool | 7-10 days
  Phase I will consist of two on line tests that assess surgical and anatomic knowledge. The tests will be separated by 7-10 days. Evaluation will determine the validity of the tests as well as creating a "knowledge curve." Analyzing resident and faculty performance with a one-way analysis of variance, with level of training as the independent variable, will assess construct validity. Post hoc contrasts are done with Student-Newman-Keuls test. We will also evaluate the validity of the exam by comparing the performance of novice surgeons with more advanced residents and experts. Internal consistency of the examination, which is a measure of the reliability of the test, will be calculated using Cronbach's alpha test. Results will be presented as percentages, means and standard deviations based on the number of questions that are answered correctly.

SECONDARY OUTCOMES:
Number of experts using validation tool | 7-10 days
  Phase I will consist of two on line tests that assess surgical and anatomic knowledge. The tests will be separated by 7-10 days. Evaluation will determine the validity of the tests as well as creating a "knowledge curve." Analyzing resident and faculty performance with a one-way analysis of variance, with level of training as the independent variable, will assess construct validity. Post hoc contrasts are done with Student-Newman-Keuls test. We will also evaluate the validity of the exam by comparing the performance of novice surgeons with more advanced residents and experts. Internal consistency of the examination, which is a measure of the reliability of the test, will be calculated using Cronbach's alpha test. Results will be presented as percentages, means and standard deviations based on the number of questions that are answered correctly.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Satkunaratnam Abheha, MD, Principal Investigator — Unity Health Toronto
Locations (6):
- United States (3):
  - University of Southern California, Department of Obstetrics and Gynecology, Los Angeles, California
  - University of California Los Angeles, Department of Obstetrics and Gynecology, Los Angeles, California
  - University of Washington, School of Medicine, Department of Obstetrics and Gynecology, Seattle, Washington
- Canada (2):
  - University of British Columbia, Division of Obstetrics and Gynecology, Vancouver, British Columbia
  - University of Toronto Faculty of Medicine, Toronto, Ontario
- University Medical Center, Utrecht, The Netherlands, Utrecht, Heidelberglaan, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided